CLINICAL TRIAL: NCT01256060
Title: Intranasal Oxytocin for the Treatment of Children and Adolescents With Autism Spectrum Disorders (ASD)
Brief Title: Intranasal Oxytocin for the Treatment of Children and Adolescents With ASD (OXY)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evdokia Anagnostou (Individual)
Collaborators: Holland Bloorview Kids Rehabilitation Hospital (Other); The Hospital for Sick Children (Other); University of Illinois at Chicago (Other)
Responsible Party: Sponsor-Investigator, Evdokia Anagnostou, Principal Investigator, Anagnostou, Evdokia, M.D.
Organization: Anagnostou, Evdokia, M.D. (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-001
Record Dates: First submitted 2010-11-22; First posted 2010-12-08 (Estimated); Results first posted 2015-04-15 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum disorder; Oxytocin; Clinical Trial; Children; Pharmacology
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intanasal Oxytocin (Experimental): A modified dose finding method will be used to determine safety among four dose levels for Intranasal Oxytocin. Half the dose (0.2 IU/kg /dose) is the minimum dose and two intermediate doses will also be evaluated (0.26 and 0.33 IU/kg / dose) Dose-finding escalations will be done in groups of three patients.Three patients will be studied at the first dose level. If none of these patients experience dose limiting toxicity, the dose will be escalated. If one experiences dose limiting toxicity, up to three more will be accrued at the same level. If none of these experience dose limiting toxicity, the dose will be escalated. If one or more of these experience dose-limiting toxicity, entry at that dose level will be stopped. Up to three more patients will be treated at the next lower dose. If zero out of these experience dose limiting toxicity, an additional three patients will be treated at that dose.
  Interventions: Drug: Intranasal Oxytocin

INTERVENTIONS:
Drug: Intranasal Oxytocin — We are selecting morning and afternoon dosing to try to influence most hours where youth are in settings with increased potential for social interaction (school, after school). Medication will be administered by the parents before school and early afternoon. All patients will receive their first dose by the study physician to educate parents and themselves on proper administration and determine safety of first dose.
  Other Names: Syntocinon

SUMMARY:
Extensive data has been accumulated to suggest that central release of oxytocin is important for social cognition and function, as well as likely involved in anxiety modulation and repetitive behaviors. The principal investigators of this study have previously documented: 1) an association between Autism Spectrum Disorder and a single nuclear polymorphism of the oxytocin receptor gene, 2) ability to measure oxytocin levels in the blood by enzyme immunoassay and 3) preliminary data to support safety and efficacy of intranasal oxytocin in the treatment of social deficits and repetitive behaviors in adults with autism. A medication treatment targeting the core deficits of Autism Spectrum Disorder in childhood is highly valuable because it could influence the developmental trajectory and make further psychosocial interventions possible. In this context, we propose a small dose finding study to confirm that the dose used in the adult study is not more than the maximum tolerated dose in youth. '

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 10-17 years of age inclusive.
2. Meet Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision criteria for Autistic Disorder or Asperger's Disorder as established by a clinician and supported by the Autism Diagnostic Observation Schedule and the Autism Diagnostic Interview - Revised.
3. Have a Clinician's Global Impression-Severity score ≥ 4 (moderately ill) at Baseline.
4. Verbal Intelligent Quotient >/= 70.
5. If already receiving stable pharmacological and or non-pharmacologic educational, behavioral, and/or dietary interventions, have continuous participation during the preceding 3 months prior to Screening and will not electively initiate new or modify ongoing interventions for the duration of the study.
6. Have normal physical examination and laboratory test results at Screening. If abnormal, the finding(s) must be deemed clinically insignificant by the Investigator.
7. The participant and caregiver must be able to speak and understand English sufficiently to allow for the completion of all study assessments.

Exclusion Criteria:

1. Patients born prior to 35 weeks gestational age.
2. Patients with any primary psychiatric diagnosis other than autism at Screening.
3. Patients with current neurological disease, including, but not limited to, epilepsy/seizure disorder (except simple febrile seizures), movement disorder, tuberous sclerosis, fragile X, and any other known genetic syndromes, or known abnormal MRI/structural lesion of the brain.
4. Pregnant female patients, sexually active female patients on hormonal birth control and sexually active females who do not use two types of non-hormonal birth control
5. Patients with a medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. Patients with evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease.
6. Patients who are sensitive to Syntocinon or any components of its formulation
7. Patients with one or more of the following: HIV, Hepatitis B virus, Hepatitis C virus, hemophilia (bleeding problems, recent nose and brain injuries), abnormal blood pressure (hypotension or hypertension), drug abuse, immunity disorder or severe depression.
8. Patients unable to tolerate venipuncture procedures for blood sampling.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, M.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Suma Jacob, M.D., Ph.D., Principal Investigator — University of Illinois at Chicago; Jessica Brian, Ph.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Wendy Roberts, M.D., Principal Investigator — The Hospital for Sick Children; Sharon Smile, M.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Edwin Cook, M.D., Principal Investigator — University of Illinois at Chicago; Annie Dupuis, Ph.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Margot Taylor, Ph.D., Principal Investigator — The Hospital for Sick Children
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the hospital clinical database, as well as presentations at local conferences and media. Diagnosis was established using the Diagnostic and Statistical Manual, Fourth Edition for an Autism Spectrum Disorder supported by the Autism Diagnostic Observations Schedule and the Autism Diagnostic Interview - Revised.
Pre-assignment Details: Cohort 1 Dosage: 0.20 IU/kg - 3 participants Cohort 2 Dosage: 0.26 IU/kg - 3 participants Cohort 3 Dosage: 0.33 IU/kg - 3 participants Cohort 4 Dosage: 0.40 IU/kg - 6 participants
Period: Overall Study
Arm/Group | 0.2 IU / kg | 0.26 IU / kg | 0.33 IU / kg | 0.4 IU / kg
Started | 3 | 3 | 3 | 6
Completed | 3 | 2 | 3 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intanasal Oxytocin: A modified dose finding method was used to determine safety among four dose levels. Half the dose (0.2 IU/kg /dose) was the minimum dose and two intermediate doses were also evaluated (0.26 and 0.33 IU/kg / dose) Dose-finding escalations were done in groups of three patients.
  1. Three patients were studied at the first dose level
  2. If none of these patients experienced dose limiting toxicity, the dose was escalated.
  3. If one patient experienced dose limiting toxicity, up to three more patients were accrued at the same level. (a) If none of these patients experienced dose limiting toxicity, the dose was escalated. (b) If one or more experienced dose-limiting toxicity, entry at that dose level would be stopped, the maximum tolerated dose exceeded, and dose escalation would be stopped. Up to three more patients would be treated at the next lower dose. If zero out of three patients experience dose limiting toxicity, an additional three patients were to be treated at that dose.
Arm/Group | Intanasal Oxytocin
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Region of Enrollment [Number; unit: participants]
  Canada | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The hypothesis is that the maximum tolerated dose in a range of 0.2-0.4 IU/kg / dose will be 0.4 IU/kg / dose, as was the case in the adult study, given that oxytocin is not stored in body fat and does not depend on liver or renal clearance.
Time Frame: 12 Weeks
Measure: Number; unit: IU / kg
Groups:
- Intanasal Oxytocin: Cohort 1 Dosage: 0.20 IU/kg - 3 participants Cohort 2 Dosage: 0.26 IU/kg - 3 participants Cohort 3 Dosage: 0.33 IU/kg - 3 participants Cohort 4 Dosage: 0.40 IU/kg - 6 participants
Arm/Group | Intanasal Oxytocin
Number analyzed (Participants) | 15
IU / kg | 0.40

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: This will be reported as the number of participants who experienced a serious advert event throughout the study.
Time Frame: 24 Weeks
Measure: Number; unit: participants
Groups:
- Intanasal Oxytocin: Number of Participants Experiencing a Serious Adverse Event
Arm/Group | Intanasal Oxytocin
Number analyzed (Participants) | 15
participants | 0

3. Secondary Outcome: Baseline Levels of Oxytocin in Relation to Either Safety or Treatment Response
Description: Children and adolescents with lower plasma oxytocin levels at baseline will show treatment related changes in social cognition. Children and adolescents with higher oxytocin plasma levels will show diminished or less dramatic treatment responses and may have more difficulty tolerating the treatment.
Time Frame: 12 Weeks
Reporting Status: Not Posted, anticipated posting 2016-12

4. Secondary Outcome: Blood Levels of Oxytocin During the Trial in Relation to Safety or Treatment Response
Description: Children and adolescents with minimal changes in plasma level of oxytocin after treatment will be less responsive to treatment. Children and adolescents with atypical patterns of increase in oxytocin may be more sensitive to dose-related tolerability.
Time Frame: 12 Weeks
Reporting Status: Not Posted, anticipated posting 2016-12

5. Other Pre Specified Outcome: Changes in Measures of Social Cognition, Social Function, Repetitive Behaviors, and Anxiety (Baseline to Week 12)
Description: Social Cognition (higher score=positive response)
  1. Let's Face It Skills Battery; i. Matchmaker (0-100); ii. Faces (0-100); iii. Houses (0-100)
  2. Eyes Test (0-28)
  3. Strange Stories (0-16)
  4. Irony and Empathy (0-24)
  Social Function
  1. Aberrant Behavior Checklist (0-48) (lower score=positive response)
  2. Behavioral Assessment System for Children (higher score=positive response); i. Social: age 8 to 11 & 15 to 18 (18-69); age 12 to 14 (21-70); ii. Functional: age 8 to 14 (10-66); age 15 to 18 (10-64)
  3. Social Responsiveness Scale (higher score=positive response); male (34-127); female (35-142)
  Anxiety (lower score=positive response)
  a. Child Symptom Inventory; i. Separation: male (44-106); female (44-101); ii. Generalized: male (40-101); female (41-96)
  Repetitive Behaviors (lower score=positive response)
  1. Child Yale-Brown Obsessive-Compulsive Scale (0-20)
  2. Repetitive Behavior Scale (0-129)
  Measures insensitive to change will be omitted from results.
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intranasal Oxytocin: Oxytocin: Intranasal Oxytocin
Arm/Group | Intranasal Oxytocin
Number analyzed (Participants) | 15
units on a scale
  Let's Face It! Skills Battery-Matchmaker | -10.9 [-19.3 to -2.6]
  Let's Face It! Skills Battery-Faces | -9.21 [-15.26 to -3.15]
  Let's Face It! Skills Battery-Houses | -10.73 [-18.5 to -2.91]
  The Revised Eyes Test | -0.14 [-0.82 to 0.53]
  Strange Stories Task | -1.36 [-2.72 to 0.0008]
  Irony and Empathy Task | -1.64 [-3.02 to -0.27]
  Aberrant Behavior Checklist | 3.00 [0.05 to 5.96]
  Social Responsiveness Scale | 9.8 [3.8 to 15.8]
  Behavioral Assessment System for Children-Social | -2.84 [-5.31 to -0.38]
  Behavioral Assessment System for Children-Function | -4.10 [-6.23 to -1.97]
  Child Yale-Brown Obsessive-Compulsive Scale | 2.93 [0.95 to 4.91]
  Repetitive Behavior Scale-Revised | 17.3 [6.3 to 28.3]
  Child and Adolescent Symptom Inventory-Separation | 7.5 [0.2 to 14.8]
  Child and Adolescent Symptom Inventory-General | 11.0 [4.0 to 18.0]

6. Other Pre Specified Outcome: Measures of Social Function - The Clinical Global Impressions - Social Scale (Baseline to Week 12)
Description: Social Function
  a) Clinical Global Impressions - Social Scale (1-7) (lower score=positive response). The results will be reported as the number of participants that were classified as a social responder (achieving a score of 1 or 2 on the scale).
Time Frame: 12 Weeks
Measure: Number; unit: participants
Arm/Group | Intranasal Oxytocin
Number analyzed (Participants) | 15
participants | 7

ADVERSE EVENTS:
Groups:
- Intranasal Oxytocin: Oxytocin: Intranasal Oxytocin. Please note that the Adverse Events are not presented per dose level received, as this is not a dose-finding study, it is a modified maximum tolerated dose study. This means that a small number of participants were exposed to increasing dose levels to assess for Adverse Events. It is not meaningful to analyze adverse events by cohorts due to the extremely small sample size.
Arm/Group | Intranasal Oxytocin
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Oxytocin (N=15)
Emotional Lability (Nervous system disorders) | 6 (7)
Irritability (Psychiatric disorders) | 4 (6)
Headache (Nervous system disorders) | 7 (11)
Migraine (Nervous system disorders) | 1 (3)
Abdominal Discomfort (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (2)
Upper Respiratory Infections (Infections and infestations) | 6 (7)
Decrease Appetite (Metabolism and nutrition disorders) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Itchy Nose (Skin and subcutaneous tissue disorders) | 1 (2)
Fatigue (General disorders) | 4 (5)
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Tooth Sensitivity/Pain (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The sample size is too small to view both safety and efficacy data. The design did not exceed the commonly used 24 IU / dose, so it is not clear that higher doses would not confer benefit. In the absence of placebo, adverse events may be inflated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No